CLINICAL TRIAL: NCT00541827
Title: Skeletal Muscle and Platelet Mitochondrial Dysfunction During Sepsis
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: assente
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Sepsis. Shock, septic. Mitochondria.
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — muscle tissue, platelets, plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary aim of the study is to demonstrate that mitochondrial dysfunction occurs in both skeletal muscle and circulating platelets of severely septic and septic shock ICU-admitted patients. Secondary aims are to clarify the pathogenesis and the clinical relevance of mitochondrial damage during sepsis.

DETAILED DESCRIPTION:
The primary aim of the study is to demonstrate that mitochondrial dysfunction occurs in both skeletal muscle and circulating platelets of severely septic and septic shock ICU-admitted patients, as compared to otherwise healthy surgical ones. In order to better clarify the pathogenesis of mitochondrial dysfunction during sepsis, cardiogenic shock patients (suffering from systemic hypoperfusion) will act as additional controls. Markers of oxidative stress will be measured in tissue samples from septic patients. The clinical relevance of mitochondrial dysfunction during sepsis will be assessed in terms of both skeletal muscle and platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive ICU-admitted severely septic or septic shock patients.

Exclusion Criteria:

* Severe thrombocytopenia.
* Severe coagulopathy.
* Pre-existing mitochondrial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult ICU-admitted severely septic and septic shock patientes; adult ICU-admitted cardiogenic shock patients; surgical patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Mitochondrial respiratory chain enzyme activity | On day one and seven from admission to ICU

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Gattinoni, MD, Study Chair — Ospedale Maggiore Policlinico Mangiagalli e Regina Elena; Alessandro Protti, MD, Principal Investigator — Ospedale Maggiore Policlinico Mangiagalli e Regina Elena
Locations (1):
- Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan, Italy, Italy

REFERENCES:
- [Derived] Protti A, Fortunato F, Artoni A, Lecchi A, Motta G, Mistraletti G, Novembrino C, Comi GP, Gattinoni L. Platelet mitochondrial dysfunction in critically ill patients: comparison between sepsis and cardiogenic shock. Crit Care. 2015 Feb 11;19(1):39. doi: 10.1186/s13054-015-0762-7. PMID 25757508